CLINICAL TRIAL: NCT01011140
Title: Physician Perceptions About Parenteral Hydration in Latin America and Spain: A Survey of Physicians Affiliated With the Latin American Association for Palliative Care (ALCP) and the Spanish Society for Palliative Care (SECPAL)
Brief Title: Physician Perceptions About Parenteral Hydration in Latin America and Spain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0606
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Dehydration; Advanced Cancers
Keywords: Parenteral Hydration; Latin American Association for Palliative Care; ALCP; Spanish Society for Palliative Care; SECPAL; Online survey; Palliative care; Physicians' attitudes; End of life; Latin America; Spain
MeSH Terms: conditions — Dehydration; Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Online Survey: Survey of Palliative care physicians from Latin America and Spain
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — 10-15 minute online survey to assess palliative care physicians' attitudes, beliefs and practice patterns related to parenteral hydration at the end of life in Latin America and Spain.
  Other Names: Questionnaire

SUMMARY:
The purpose of this study is to assess palliative care physicians' attitudes, beliefs and practice patterns related to parenteral hydration at the end of life in Latin America and Spain.

Objectives:

1. To assess palliative care physicians' attitudes, beliefs and practice patterns related to parenteral hydration at the end of life in Latin America and Spain.
2. To assess cross-national differences in practice patterns related to parenteral hydration at the end of life. (Latin America vs. Spain).
3. To determine the percentage of physicians who practice parenteral hydration at the end-of-life in the hospital setting and the home setting.
4. To examine the association between providers' parenteral hydration practice patterns and:

   * 1. provider demographic characteristics;
   * 2. specific characteristics of their practice settings; and
   * 3. training and experience in end of life care;
5. To determine which factors most predict the practice of parenteral hydration at the end of life among palliative care physicians.

DETAILED DESCRIPTION:
This study is a collaboration between MD Anderson's Departments of Palliative care and Rehabilitation Medicine, Health Disparities Research, the Latin American Association for Palliative Care (ALCP) and the Spanish Society for Palliative Care (SECPAL). The proposed study involves a 10-15 minute online survey of palliative care physicians from Latin America and Spain to assess their attitudes, beliefs and practice patterns related to parenteral hydration at the end of life.

ELIGIBILITY:
Inclusion Criteria:

1. Palliative care physicians practicing in Latin America and Spain and affiliated with either the ALCP or SECPAL.
2. Physicians must report dedicating at least 30% of their practice to palliative care.
3. Physician must be 18 years of age or older.

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians affiliated with the Latin American Association for Palliative Care (ALCP) and the Spanish Society for Palliative Care (SECPAL)
Sampling Method: Non-Probability Sample
Enrollment: 516 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of terminally ill cancer patients overall that receive an order of parenteral hydration as reported by physicians | Online Survey, completion any time during estimated 2 month period

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Torres, MPH, DRPH, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org